CLINICAL TRIAL: NCT07101406
Title: The Effect of TUBER Recommendations and the DASH Diet on Blood Parameters in Patients With Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kardelen Kandemir (Other)
Responsible Party: Sponsor-Investigator, Kardelen Kandemir, Research Asisstant (Dietitian), Atlas University
Organization: Atlas University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 28.06.2024-993310
Record Dates: First submitted 2025-07-24; First posted 2025-08-03 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Gestational Diabetes Mellitus (GDM); Gestational Diabetes Mellitus in Pregnancy, Diet- Controlled
Keywords: gestational diabetes; dash diet; Türkiye Nutrition Guide; diet
MeSH Terms: conditions — Diabetes, Gestational | interventions — Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Intervention Model Description: Randomized single-blind. Participants were blinded.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: Türkiye Nutrition Guideline Diet Group (Active Comparator): Participants followed a diet based on the Türkiye Nutrition Guideline (TÜBER) for pregnancy. The diet consisted of 45-60% carbohydrates, 12-20% protein (minimum 70 g), and 20-35% fat. Portion sizes were explained during the initial consultation. Participants recorded their food intake weekly and attended weekly follow-up visits for anthropometric and blood pressure measurements. Diets were adjusted weekly based on blood glucose levels.
  Interventions: Other: Türkiye Nutrition Guideline Diet
- Active Comparator: DASH Diet Group (Active Comparator): Participants followed a diet based on the Dietary Approaches to Stop Hypertension (DASH) guidelines. The diet consisted of 45-60% carbohydrates (minimum 175 g), 12-20% protein (minimum 70 g), and 20-35% fat including 6% saturated fat and 150 mg cholesterol. It was low in sodium (2300 mg/day) and rich in potassium (4700 mg), calcium (1250 mg), and magnesium (500 mg). It emphasized low-fat dairy, lean meats, 10 servings/day of fruits and vegetables, and 4-5 servings/week of nuts, seeds, and legumes. Weekly follow-ups were conducted as in the other group.
  Interventions: Other: DASH Diet

INTERVENTIONS:
Other: Türkiye Nutrition Guideline Diet — A diet structured according to the Türkiye Nutrition Guideline (TÜBER) for pregnant women, consisting of 45-60% carbohydrates, 12-20% protein (minimum 70 g), and 20-35% fat. Diets were tailored weekly based on blood glucose levels and individual dietary intake records.
  Arms: Active Comparator: Türkiye Nutrition Guideline Diet Group
Other: DASH Diet — A dietary plan based on DASH guidelines: 45-60% carbohydrates (≥175 g), 12-20% protein (≥70 g), 20-35% fat (≤6% saturated), ≤2300 mg sodium, ≥4700 mg potassium, ≥1250 mg calcium, ≥500 mg magnesium. Includes low-fat dairy, lean meats, fruits/vegetables, and nuts/seeds.
  Arms: Active Comparator: DASH Diet Group

SUMMARY:
The aim of this clinical trial was to examine the effects of the Turkish Nutrition Guide Recommendations Diet and the DASH Diet on blood sugar, blood pressure, and biochemical parameters in patients with gestational diabetes. The study hypotheses are as follows:

Hypothesis 1: The DASH diet reduces fasting blood glucose levels more in patients with gestational diabetes compared to a diet adapted to a healthy diet specific to Türkiye.

Hypothesis 1: The DASH diet reduces insulin levels more in patients with gestational diabetes compared to a diet adapted to a healthy diet specific to Turkey.

Hypothesis 1: The DASH diet reduces HbA1c levels more in patients with gestational diabetes compared to a diet adapted to a healthy diet specific to Türkiye.

Hypothesis 1: The Dash diet reduces 1st-hour postprandial glucose levels more significantly in women with gestational diabetes compared to a diet adapted to a healthy diet typical of Türkiye.

Participants:

After being diagnosed with gestational diabetes by a doctor using an OGTT test at 24-28 weeks, the researcher will complete a general information form during their first consultation with the dietitian. For four weeks, the dietitian will follow the diets created by the researcher based on their assigned diet group in a blinded manner. They will record their fasting and postprandial blood sugar levels in the morning, noon, evening, night, and during snacks, if they are taking them. They will keep a 24-hour food consumption record before meeting with the researcher weekly. Participants will have their biochemical parameters assessed at the beginning of the study and at the end of the fourth week.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18 to 35 years
* Singleton pregnancy
* Clinical diagnosis of gestational diabetes mellitus (GDM)
* Ability to use a glucometer

Exclusion Criteria:

* Pre-gestational diabetes or impaired glucose tolerance (IGT)
* Hypoglycemia
* Receiving insulin therapy
* Development of preeclampsia
* Failure to adhere to the prescribed diet
* Smoking
* Alcohol consumption

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 38 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Change in fasting blood glucose levels | Daily for 4 weeks
  To monitor daily fasting blood glucose levels (mg/dL) using a glucometer throughout the 4-week intervention.

SECONDARY OUTCOMES:
Change in 1-hour postprandial blood glucose levels | Daily for 4 weeks
  To track 1-hour post-meal blood glucose levels (mg/dL) recorded daily throughout the study.
Change in fasting insulin level | Baseline and Week 4
  To evaluate changes in fasting insulin levels (µIU/mL) from baseline to the end of the 4-week intervention period.
Change in daily energy and nutrient intake based on 24-Hour Food Consumption Record | Baseline and weekly over 4 weeks
  To assess participants' dietary intake patterns and nutrient adequacy by analyzing the 24-Hour Food Consumption Record collected at baseline and during follow-up. The analysis includes total daily energy intake (kcal) and macronutrient (carbohydrates, protein, fat) and micronutrient (iron, folic acid, vitamin D, etc.) intake levels.
  Energy: kcal/day
  Macronutrients: grams/day (carbohydrates, protein, fat)
  Micronutrients: mg or µg/day (iron, folic acid, vitamin D, etc.)
Change in lipid profile (total cholesterol, HDL-C, LDL-C, triglycerides) | Baseline and Week 4
  To evaluate the effect of the dietary intervention on lipid metabolism by measuring changes in total cholesterol, HDL cholesterol, LDL cholesterol (direct measurement), and triglyceride levels from baseline to week 4. Each parameter will be analyzed individually and reported in mg/dL.
  Total cholesterol (mg/dL)
  HDL cholesterol (mg/dL)
  LDL cholesterol - direct measurement (mg/dL)
  Triglycerides (mg/dL)
Change in iron-related parameters (iron, ferritin, total iron-binding capacity) | Baseline and Week 4
  To assess the effect of the intervention on iron status by measuring serum iron, ferritin, and total iron-binding capacity (TIBC) at baseline and Week 4.
  Iron: mcg/dL
  Ferritin: mcg/L
  TIBC: mcg/dL
Change in vitamin and hematological markers (Vitamin D, folic acid, hemoglobin, hematocrit) | Baseline and Week 4
  To evaluate changes in nutritional and hematological status from baseline to the end of the intervention period.
  25-OH vitamin D: mcg/L
  Folic acid: mcg/dL
  Hemoglobin: g/dL
  Hematocrit: %
Change in HbA1c level | Baseline and Week 4
  To assess the effect of the dietary intervention on long-term glycemic control by measuring HbA1c levels (%) before and after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Atlas Univercity Hospital, Istanbul, Bagcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided